CLINICAL TRIAL: NCT02214680
Title: The Effect of Topical Treatment With Combigan Compared to Timolol and Brimonidine on Pupil Diameter
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Orna Geyer, Professor, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CMC-14-0016-CTIL; CMC-14-0016 (Other: Carmel Medical Center)
Record Dates: First submitted 2014-08-11; First posted 2014-08-12 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Pupil diameter; Brimonidine; Timolol; Combigan
MeSH Terms: interventions — Brimonidine Tartrate, Timolol Maleate Drug Combination; Timolol; Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination of Brimonidine and Timolol (Experimental): On the first exam the subject will receive Combigan (Combination of Brimonidine and Timolol) eye drop to the right eye and a Brimonidine drop to the left eye. The effect on pupil size before and 30 minutes, 60 minutes, 240 minutes, and 300 minutes after instillation of eyedrops. On the second exam the subject will receive Timolol (0.5%) eye drop to the right eye and a Brimonidine drop to the left eye. The effect on pupil size before and 30 minutes, 60 minutes, 240 minutes, and 300 minutes after instillation of eyedrops.
  Interventions: Drug: Combigan (Combination of Brimonidine and Timolol); Drug: Timolol

INTERVENTIONS:
Drug: Combigan (Combination of Brimonidine and Timolol) — On the first exam the subject will receive Combigan (Combination of Brimonidine and Timolol) eye drop to the right eye and a Brimonidine drop to the left eye. The effect on pupil size before and 30 minutes, 60 minutes, 240 minutes, and 300 minutes after instillation of eyedrops. On the second exam the subject will receive Timolol (0.5%) eye drop to the right eye and a Brimonidine drop to the left eye. The effect on pupil size before and 30 minutes, 60 minutes, 240 minutes, and 300 minutes after instillation of eyedrops.
  Other Names: Alphagan; Tiloptic; Combigan
Drug: Timolol — 0.5% eye drop
  Other Names: Tiloptic

SUMMARY:
In this study we will explore the combined effect of Brimonidine and Timolol 0.5% (Combigan) eye drops on pupil dilation. It is a well studied phenoma that Brimonidine and a miotic effect on the pupil, however the combined effect of alpha agonist and beta blocker has not been studied.

DETAILED DESCRIPTION:
In this study we will explore the combined effect of Brimonidine and Timolol 0.5% (Combigan) eye drops on pupil dilation. It is a well studied phenoma that Brimonidine and a miotic effect on the pupil, however the combined effect of alpha agonist and beta blocker has not been studied.

The study subjects will be examined twice, two weeks apart. On the first exam the subject will receive Combigan eye drop to the right eye and a Brimonidine drop to the left eye. The effect on pupil size before and 30 minutes, 60 minutes, 240 minutes, and 300 minutes after instillation of eyedrops. On the second exam the subject will receive Timolol (0.5%) eye drop to the right eye and a Brimonidine drop to the left eye. The effect on pupil size before and 30 minutes, 60 minutes, 240 minutes, and 300 minutes after instillation of eyedrops.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults subjects with no ocular pathology
* Non pregnant women
* Normal pupil response

Exclusion Criteria:

* Chronic topical treatment
* Systemic medication affecting autonomic nerve system
* History of intra-ocular surgery
* Irregular pupil
* History of ocular neurological or severe cardio-vascular disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pupil diameter | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Orna Geyer, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel